CLINICAL TRIAL: NCT02687217
Title: Role of Perioperative Hyperoxygenation in Wound Infection Following Surgery for Acute Appendicitis: A Randomised Controlled Trial.
Brief Title: Effect of Peri-operative Supplemental Oxygen in Wound Infection After Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Swati Sattavan, Senior Resident, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LHMC/ECHR/2014/326
Record Dates: First submitted 2016-02-09; First posted 2016-02-22 (Estimated); Results first posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Perioperative Hyperoxygenation; Wound Infection
Keywords: PerioperativeHyperoxygenation; Wound Site Infection; Appendicitis
MeSH Terms: conditions — Wound Infection; Appendicitis | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: Control (No Intervention): Group A: Control- Received no supplemental oxygen throughout the surgery and received oxygen at 4l/min. in 2hrs postoperatively
- Group B: Test (Experimental): Group B: Test- Received hyperoxygenation more than or equal to 50% throughout the surgery and received oxygen at 6l/min. upto 2 hrs postoperatively.
  Interventions: Drug: oxygen

INTERVENTIONS:
Drug: oxygen — Hyperoxygenation ≥50% of oxygen by mask(non-rebreathing) was given through out the surgery.
  Received 6L/min of oxygen through venturimask upto 2 hours in post operative period.
  Hyperoxygenation refers to provision of ≥50% of oxygen by mask(non-rebreathing) through out the surgery.
  Arms: Group B: Test

SUMMARY:
The study evaluates the role of supplemental hyper-oxygenation given perioperatively on wound site infection after appendectomy. Half of the patients received ≥50% oxygen and half of them received no oxygen during the surgical procedure.

DETAILED DESCRIPTION:
Patient with the diagnosis of acute appendicitis of >15 years of age group, with no comorbidities who presented to surgical emergency in Dr. Ram Manohar Lohia Hospital were considered for the present study.

30 patients who fulfilled the inclusion criteria and who voluntarily consented for the study were randomly allocated to the two groups- Group A (control group) and Group B (study group).

These patients were operated through Mc-Burney incision given in the right lower quadrant.

Both the groups were comparable in their demographic and preoperative profile. The study group was given ≥50% of oxygen intraoperatively and the control group was given no oxygen.

In postoperative period, oxygen was given to group A at the rate of 4 litre/minute (L/min) and group B at the rate of 6 litre/minute (L/min).

The assessment of the wound was done by using ASEPSIS (Additional treatment; Serous discharge; Erythema; Purulent exudate; Separation of deep tissues; Isolation of bacteria; and Stay) score. A score of more than 20 is considered to be infected.

Fever, raised total leucocyte count, positive pus culture, Ultrasound evidence of fluid collections, removal of sutures and duration of hospital stay were also measured for the evaluation of economic implications due to SSI.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis or Radiological diagnosis of acute appendicitis.
2. Appendectomy through the Mc Burney incision.

Exclusion Criteria:

1. Patients with chronic obstructive pulmonary diseases.
2. Immunodeficiency disease.
3. Patients requiring midline incision.
4. Patients requiring general anaesthesia after failure of spinal anaesthesia.
5. Patients requiring higher oxygen in perioperative period.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Swati Sattavan, M.S., Principal Investigator — Lady Hardinge Medical College and Associated Hospitals

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B: Test: Group B: Test- Received hyperoxygenation more than or equal to 50% throughout the surgery and received oxygen at 6l/min. upto 2 hrs postoperatively.
  oxygen: Hyperoxygenation refers to provision of ≥50% of oxygen by mask(non-rebreathing) through out the surgery.
Period: Overall Study
Arm/Group | Group A: Control | Group B: Test
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Group A: Control:
  1. No supplemental oxygen throughout surgery.
  2. Received oxygen 4L/min. in 2 hrs postoperative period through venturimask.
  Group B: Test:
  1. Hyperoxygenation ≥50% of oxygen by mask(non-rebreathing) was given through out the surgery.
  2. Received 6L/min of oxygen through venturimask upto 2 hrs in post operative period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A: Control | Group B: Test | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Customized [Number; unit: participants]
  15-20 years | 7 | 8 | 15
  21-25 years | 9 | 10 | 19
  26-30 | 7 | 7 | 14
  31-35 | 3 | 2 | 5
  36-40 | 3 | 2 | 5
  41-45 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 23 | 23 | 46
Body Mass Index [Mean (Standard Deviation); unit: Kg/m^2] | 22.71 (3.17) | 23.35 (4.25) | 22.81 (3.7)
Body temperature [Mean (Standard Deviation); unit: degrees Fahrenheit] | 98.45 (1.01) | 98.67 (1.16) | 98.56 (1.08)
Abdominal pain duration [Mean (Standard Deviation); unit: days] | 1.33 (0.54) | 1.87 (0.86) | 1.60 (0.76)
Preoperative Haemoglobin [Mean (Standard Deviation); unit: g/dL] | 12.87 (1.17) | 13.07 (1.57) | 12.97 (1.38)
Preoperative Total leucocyte count [Mean (Standard Deviation); unit: 10^3 cells per mm^3] | 12.20 (1.71) | 13.30 (3.65) | 12.75 (2.88)
Haemodynamic parameter [Number; unit: participants] — Stable: With normal haemodynamic parameter. Unstable: With deranged hemodynamic parameter.
  participants
    Stable | 30 | 30 | 60
    unstable | 0 | 0 | 0
Intraoperative pH [Mean (Standard Deviation); unit: pH] | 7.39 (0.03) | 7.40 (0.05) | 7.39 (0.04)
Intraoperative partial pressure of arterial oxygen [Mean (Standard Deviation); unit: mmHg] | 86.53 (3.52) | 151.67 (2.88) | 119 (3.86)
Intraoperative partial pressure of carbon dioxide [Mean (Standard Deviation); unit: mmHg] | 36.82 (2.78) | 36.16 (6.46) | 36.49 (4.94)
Intraoperative bicarbonate [Mean (Standard Deviation); unit: mmol/L] | 23.12 (1.2) | 23.60 (3.39) | 23.36 (2.53)
Intraoperative oxygen saturation [Mean (Standard Deviation); unit: percentage of oxygenated haemoglobin] | 97.01 (5.20) | 98.50 (1.08) | 97.76 (3.80)
Intraoperative findings [Number; unit: participants]
  Acute Appendicitis | 29 | 26 | 55
  Gangrenous Appendicitis | 1 | 4 | 5
Duration of surgery [Mean (Standard Deviation); unit: Hours] | 1.05 (.15) | 1.14 (.29) | 1.1 (.23)
Postoperative partial pressure of arterial oxygen [Mean (Standard Deviation); unit: mmhg] | 86.21 (3.85) | 137.6 (2.49) | 119 (3.13)
Postoperative Total leucocyte count [Mean (Standard Deviation); unit: 10^3 cells per mm^3] | 8.16 (1.17) | 9.03 (2.10) | 8.6 (1.74)
Use of antibiotics [Mean (Standard Deviation); unit: days] | 5.26 (1.11) | 5.60 (1.27) | 5.43 (1.19)
length of hospital stay [Mean (Standard Deviation); unit: days] | 3.87 (1) | 3.87 (1) | 3.87 (1)

OUTCOME MEASURES:

1. Primary Outcome: ASEPSIS Score
Description: ASEPSIS score- Additional treatment; Serous discharge; Erythema; Purulent exudate; Separation of deep tissues; Isolation of bacteria; and Stay. A daily score of 20 or more considered evidence of infection.
  Category of infection:
  Total score of 0-10 satisfactory healing; 11-20 disturbance of healing; 21-30 minor wound infection; 31-40 moderate wound infection; > 40 severe wound infection.
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Group A: Control | Group B: Test
Number analyzed (Participants) | 30 | 30
participants
  Satisfactory healing | 30 | 30
  Disturbance of healing | 0 | 0
  Minor wound infection | 0 | 0
  Moderate wound infection | 0 | 0
  Severe wound infection | 0 | 0
Statistical Analysis 1: Comparison: Group A: Control vs Group B: Test; Test type: Superiority or Other; p = 0.5, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Patients Requiring Additional Investigations
Description: Sonography; Pus culture; blood culture; Total Leucocyte Count.
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Group A: Control | Group B: Test
Number analyzed (Participants) | 30 | 30
participants
  Required | 0 | 0
  Not required | 30 | 30
Statistical Analysis 1: Comparison: Group A: Control vs Group B: Test; Test type: Superiority or Other; p = 0.5, Chi-squared

3. Secondary Outcome: Number of Patients Requiring Additional Treatment
Description: Requirement of antipyretics; increased dose/ duration of antibiotic usage other than standard protocol; need for change to higher antibiotics; requirement of drainage procedures for pus/ wound infections; requirement for additional dressing sessions
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | Group A: Control | Group B: Test
Number analyzed (Participants) | 30 | 30
participants
  Required | 0 | 0
  Not required | 30 | 30
Statistical Analysis 1: Comparison: Group A: Control vs Group B: Test; Test type: Superiority or Other; p = 0.5, Chi-squared

ADVERSE EVENTS:
Arm/Group | Group A: Control | Group B: Test
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
The study included a small sample size of 60 patients, randomized into equal study group and control group as the time limit restrictions of 12- 15 months as prescribed by the residency programme.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes